CLINICAL TRIAL: NCT07299877
Title: Perineural Dexamethasone, Dexmedetomidine or Their Combination: an Effort to Reduces Rebound Pain After Supraclavicular Brachial Plexus Block: A Triple-Blind Randomized Controlled Trial
Brief Title: Perineural Dexamethasone, Dexmedetomidine, or Their Combination to Reduces Rebound Pain After Supraclavicular Brachial Plexus Block
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC. 10.9.2025
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Brachial Plexus Blocks
Keywords: Dexamethasone; dexmedetomidine
MeSH Terms: interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): 8 mg of dexamethasone will be added to the local anesthetic.The local anesthetic that will be used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Interventions: Drug: Group A (Dexamethasone)
- Group B (Active Comparator): 1 microgram/kg of dexmedetomidine will be added to the local anesthetic. The local anesthetic that will be used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Interventions: Drug: Group B (Dexmedetomidine)
- Group C (Active Comparator): 8 mg of dexamethasone + 1 microgram/kg of dexmedetomidine will be added to the local anesthetic. The local anesthetic that will be used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Interventions: Drug: Group C (Dexamethasone + Dexmedetomidine)

INTERVENTIONS:
Drug: Group A (Dexamethasone) — 8 mg of dexamethasone will be added to the local anesthetic. The local anesthetic used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Arms: Group A
Drug: Group B (Dexmedetomidine) — 1 microgram/kg of dexmedetomidine will be added to the local anesthetic. The local anesthetic used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Arms: Group B
Drug: Group C (Dexamethasone + Dexmedetomidine) — 8 mg of dexamethasone + 1 microgram/kg dexmedetomidine will be added to the local anesthetic. The local anesthetic used in all cases was a mixture of 10 ml of 2% xylocaine and 10 ml of 0.5% bupivacaine.
  Arms: Group C

SUMMARY:
Dexmedetomidine, an α2 adrenoceptor agonist, and dexamethasone, a potent anti-inflammatory steroid, are commonly used, effective, and safe adjuvants to peripheral nerve block (PNB). Both have been found to delay and reduce the incidence of rebound pain (RP), prolong the duration of sensory and motor block, and enhance analgesia without causing significant respiratory depression. Few studies have explored the effectiveness of dexmedetomidine or dexamethasone as sole adjuvants to PNB for preventing or reducing RP. However, no study has directly compared the effectiveness of these two drugs in reducing RP when used as adjuvants to local anesthetic (LA) in PNB. Due to differences in their mechanism of action, their effects on RP may differ significantly. The investigators hypothesized that the combination of dexamethasone and dexmedetomidine reduces the incidence of RP when used as adjuvants to LA in PNB.

ELIGIBILITY:
Inclusion Criteria:

* from 20-65 years old
* and ASA physical status I or II and III,
* and of either gender,
* who provided informed, written, and valid consent,
* were scheduled for elective orthopedic upper limb surgeries for traumatic fractures under Supraclavicular Brachial Plexus Block.

Exclusion Criteria:

* Patients with coagulopathies,
* neurological disorders,
* hypersensitivity to any of the study drugs, or
* a history of previous surgeries on the affected limb
* and those who refused to sign informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of rebound pain after the end of anesthesia | 24 hours
  The incidence of rebound pain after the end of anaesthesia will be measured. Rebound pain refers to a transient, intense increase in pain that occurs after the resolution of a peripheral nerve block. It represents the patient's perception of a sudden change from numbness to severe pain once the block wears off - often within the first 24 hours postoperatively. The Visual Analogue Scale (VAS) will be used to measure pain intensity. It consists of a 10-centimetre horizontal line, with the left end labelled "no pain" (0) and the right end labelled "worst imaginable pain" (10).

SECONDARY OUTCOMES:
Onset of Rebound Pain | 24 hours
  The onset of rebound pain is the time interval between the resolution of the peripheral nerve block and the patient's first report of significant pain. The Visual Analogue Scale (VAS) will be used to measure a patient's subjective pain intensity. It consists of a 10-centimetre horizontal line, with the left end labelled "no pain" (0) and the right end labelled "worst imaginable pain" (10).
Duration of Rebound Pain | 24 hours
  The duration of rebound pain refers to the length of time the heightened pain persists after its onset until it returns to a baseline or tolerable level with analgesic management.
Severity of Rebound Pain | 24 hours
  The severity of rebound pain is the intensity of pain experienced after block resolution, typically measured using the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) will be used to measure a patient's subjective pain intensity. It consists of a 10-centimetre horizontal line, with the left end labelled "no pain" (0) and the right end labelled "worst imaginable pain" (10).
Time to first analgesic request | 24 hours
  The time to first request for analgeseia will be measured
Incidence of sleep disturbances due to surgical site pain | 48 hours
  Sleep disturbance due to surgical site pain refers to difficulty initiating or maintaining sleep, or poor sleep quality, directly attributed to postoperative pain from the surgical site during the recovery period (usually within the first few nights after surgery).
  Assessment Method Direct Patient Questioning
  A structured interview asking:
  "Did pain at your surgical site interfere with your sleep last night?" "How many times did you wake up because of pain?" "How would you rate your sleep quality (excellent, good, fair, poor)?" A "yes" or poor sleep rating indicates sleep disturbance.
Pain score | 24 hours
  The Visual Analogue Scale (VAS) will be used to measure a patient's subjective pain intensity. It consists of a 10-centimetre horizontal line, with the left end labelled "no pain" (0) and the right end labelled "worst imaginable pain" (10).
Consumption of fentanyl | 48 hours
  the amount of of fentanyl rescue analgesia within the first 48 hours after surgery will be documented.
Patient satisfaction. | 24 hours
  Simple, structured questions will be used postoperatively:
  "How satisfied are you with your anaesthesia care?" "Were you comfortable during and after surgery?"
  Responses are rated on a Likert scale, such as:
  1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied.
  This allows calculation of the percentage of satisfied patients (scores 4-5).

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Faculty of Medicine, Banhā, Qalyubiyya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data could be shared with a reasonable request from corresponding author
Supporting Information: Study Protocol, SAP